CLINICAL TRIAL: NCT00890656
Title: Phase II Study of Augmented Hyper-CVAD in Acute Lymphoblastic Leukemia Salvage
Brief Title: Study of Augmented Hyper-CVAD in Acute Lymphoblastic Leukemia Salvage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0166
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Results first posted 2011-08-23 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; ALL; Leukemia; Hyper-CVAD
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Cyclophosphamide; Vincristine; Doxorubicin; Calcium Dobesilate; Dexamethasone; Granulocyte Colony-Stimulating Factor; Filgrastim; Methotrexate; Cytarabine; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Augmented Hyper-CVAD (Experimental): Hyper-CVAD (courses 1, 3, 5, and 7) alternated with high-dose methotrexate/ara-C (courses 2, 4, 6, and 8) administered on day 21; Hyper-CVAD = Cyclophosphamide, Vincristine, Doxorubicin, Decadron + Pegaspargase.
  Interventions: Drug: Cyclophosphamide (CTX); Drug: Vincristine; Drug: Doxorubicin; Drug: Decadron; Drug: G-CSF; Drug: Methotrexate (MTX); Drug: Ara-C; Drug: Pegaspargase

INTERVENTIONS:
Drug: Cyclophosphamide (CTX) — 300 mg/m^2 by vein (IV) over 3 hours every 12 hours for 6 doses days 1, 2, 3 of
  Other Names: Cytoxan
Drug: Vincristine — 2 mg by vein (IV) weekly for 3: Days 1, 8, 15
  Other Names: Oncovin®
Drug: Doxorubicin — 50 mg/m^2 by vein (IV) over 24 hours
  Other Names: Adriamycin®
Drug: Decadron — 80 mg by vein (IV) or by mouth (P.O.) daily days 1-4 and 15-18
  Other Names: Dexamethasone
Drug: G-CSF — 10 mcg/kg/day (rounded) by vein (IV) or under the skin (subcutaneously) within 72 ± 48 hours
  Other Names: Neupogen®
Drug: Methotrexate (MTX) — 200 mg/m2 by vein (IV) over 2 hours followed by 800 mg/m2 over 22 hours on day 1
  Other Names: Rheumatrex®
Drug: Ara-C — 3 gm/m^2 by vein (IV) over 2 hours every 12 hours for 4 doses on days 2 and 3.
  Other Names: Cytosar-U®
Drug: Pegaspargase — 2,500 units/m2 by vein (IV) on day 1 of odd courses and day 5 of even courses
  Other Names: PEG asparaginase; Oncaspar; Polyethylene Glycol Conjugated Lasparaginase-H

SUMMARY:
The goal of this clinical research study is to learn if a special combination of chemotherapy drugs called "augmented hyper-CVAD chemotherapy" given over 6 to 8 months followed by monthly maintenance chemotherapy for one year can help to control acute lymphoblastic leukemia or lymphoblastic lymphoma. The safety of this therapy will also be studied.

DETAILED DESCRIPTION:
The augmented hyper-CVAD chemotherapy is a combination of chemotherapy drugs including cyclophosphamide, vincristine, adriamycin, dexamethasone, and pegaspargase given together for one "course" of treatment. It is called "augmented" because additional drugs are being added to the hyper-CVAD combination, which is the standard combination of chemotherapy drugs for the treatment of acute lymphoblastic leukemia or lymphoblastic lymphoma. This switches back and forth with a course of the chemotherapy drugs methotrexate and ara-C (also with vincristine, dexamethasone, and pegaspargase).

Before treatment starts, you will have a physical exam, including blood (about 8 teaspoons) tests. You will also have a bone marrow sample taken; the sample will be taken through a large needle in the hipbone.

All participants will receive 2 kinds of chemotherapy courses for a total of 8 courses. Chemotherapy courses will be given through a large vein by a central venous catheter (a plastic tube usually placed under the collarbone).

During treatment, you will have a physical exam and give blood samples (about 1 tablespoon each) at least twice a week. A bone marrow sample will be repeated 2-3 weeks after the start of treatment to check the response, and later as needed.

Course 1 will include cyclophosphamide given by vein over 2-3 hours every 12 hours. This will be given for 6 doses over 3 days (Days 1, 2 and 3). Adriamycin will be given by vein over 24 hours on Day 4. Vincristine will be given by vein over 15 to 30 minutes on Days 1, 8, and 15. Dexamethasone (a steroid) will be given by mouth or by vein on Days 1 to 4 and 15-18. Pegaspargase will be given by vein over 1-2 hours on Day 1.

G-CSF (growth colony stimulating factor) will be given starting 24 hours after each course of chemotherapy is finished (Day 5 or 6). It is given to help with rapid recovery of the normal bone marrow. G-CSF will be injected by vein or under the skin until the blood counts recover.

Treatment to the brain will be given inside the spinal fluid (spinal tap) with ara-C and methotrexate on Days 2 and 7 of Courses 1 and 2 for a total of 4 treatments. This is done to decrease the risk that the leukemia will develop there.

During Course 2, you will receive methotrexate by infusion over 24 hours on the first day and ara-C by vein at a high dose over 2 hours every 12 hours for 4 doses (Days 2 and 3). You will also receive vincristine (Days 1, 8, and 15), dexamethasone (Days 1-4 and 15-18), and pegaspargase (Day 5).

Citrovorum factor (leucovorin), an antidote for side effects of methotrexate, will be given by vein or by mouth for 2-3 days (Day 2 and on). G-CSF will be given as in Course 1 (24 hours after the chemotherapy is finished). The treatment to the brain inside the spinal fluid will be given as in Course 1 on Days 2 and 7.

The schedule of chemotherapy will switch between hyper-CVAD (Courses 3, 5, and 7) and methotrexate/ara-C (Courses 4, 6 and 8) to complete a total of 8 courses. After the 8 courses, you will go on maintenance chemotherapy. This includes daily 6-mercaptopurine taken by mouth, weekly methotrexate by vein or mouth, monthly vincristine by vein, and prednisone by mouth for 5 days every month. Maintenance therapy will continue for one year.

Treatment will be given on an inpatient or outpatient basis for the 8 intensive courses of chemotherapy, as indicated by your condition. The maintenance treatments may be given as an outpatient. Patients will be taken off study if the disease gets worse or if intolerable side effects occur.

This is an investigational study. All of the drugs are commercially available. Their use together in this study is investigational. About 90 patients will take part in this study. All will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated acute lymphoblastic leukemia (ALL) (including Burkitt's lymphoma) or lymphoblastic lymphoma in relapse or primary refractory;
* No age restrictions;
* Zubrod performance status </= 3;
* Adequate liver (bilirubin </= 3mg/dl unless considered due to tumor) and renal function (creatinine </= 3mg/dl unless considered due to tumor);
* Adequate cardiac function (New York Heart Association (NYHA) < III as assessed by history and physical examination)

Exclusion Criteria:

* Not Applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2003-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan F. Faderl, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 6/9/2003 to 10/12/2009. All patients registered at The University of Texas M.D. Anderson Cancer Center.
Period: Overall Study
Arm/Group | Augmented Hyper-CVAD
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Augmented Hyper-CVAD
Number analyzed (Participants) | 90
Age Continuous [Median (Full Range); unit: years] | 34 [14 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 50
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Remission
Description: Complete remission (CR) required a marrow with ≤ 5% blasts in a normo- or hypercellular marrow with an absolute neutrophil count (ANC) of ≥ 1 * 10^9/L and a platelet count of ≥ 100 * 10^9/L with complete resolution of all sites of extramedullary disease required.
Time Frame: Response evaluated following first course at 14 -21 days and 1-2 weeks later to confirm response status (or at the time of hematologic recovery) and with visits every 2-3 courses.
Measure: Number; unit: Participants
Arm/Group | Augmented Hyper-CVAD
Number analyzed (Participants) | 90
Participants | 41

ADVERSE EVENTS:
Time Frame: 7 years, 7 months
Arm/Group | Augmented Hyper-CVAD
Serious Adverse Events (participants affected / at risk) | 33/90
Other Adverse Events (participants affected / at risk) | 57/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Augmented Hyper-CVAD (N=90)
Neutropenic fever (Infections and infestations) | 8 (8)
Death (General disorders) | 9 (9)
Infection (Infections and infestations) | 21 (21)
Pain (General disorders) | 6 (6)
Cardiac other (Cardiac disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Allergic reaction (General disorders) | 2 (2)
Hypotension (Cardiac disorders) | 13 (13)
Syncope (Nervous system disorders) | 1 (1)
Visual loss (Eye disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fever (General disorders) | 4 (4)
GI hemmorrhage (Gastrointestinal disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Augmented Hyper-CVAD (N=90)
Nausea/Vomiting (Gastrointestinal disorders) | 32 (32)
Diarrhea (Gastrointestinal disorders) | 23 (23)
Neuropathy (Nervous system disorders) | 13 (13)
hyperglycemia (Endocrine disorders) | 17 (17)
Elevated liver function tests (Hepatobiliary disorders) | 29 (29)
Pain (General disorders) | 5 (5)
Mucositis (Gastrointestinal disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes